CLINICAL TRIAL: NCT05958745
Title: Comparison of the Effects of Green Exercise Programs Including Resistance and Aerobic Exercises on Senior Fitness, Aerobic Capacity, Intrinsic Capacity at Nursing Homes
Brief Title: Comparison of the Effects of Green Exercise Programs Including Resistance and Aerobic Exercises
Acronym: GREENCITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GREENCITY
Record Dates: First submitted 2023-06-23; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Physical Inactivity
Keywords: Physical activity; Green exercise; Elderly
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise (Experimental): 12 week aerobic exercise
  Interventions: Behavioral: Aerobic Exercise
- Aerobic + Resistance Exercise (Active Comparator): 12 week aerobic + resistance exercise
  Interventions: Behavioral: Aerobic + resistance exercise
- Control (No Intervention): control

INTERVENTIONS:
Behavioral: Aerobic Exercise — Aerobic exercise training Program
  Arms: Aerobic Exercise
Behavioral: Aerobic + resistance exercise — Aerobic + resistance exercise training Program
  Arms: Aerobic + Resistance Exercise

SUMMARY:
It was aimed to evaluate the effects of aerobic exercise and resistance exercises performed together with aerobic exercise, applied in the concept of green exercise with a multidisciplinary team (specialist doctors physiotherapists, nurses) on senior fitness, aerobic capacity and IC in individuals aged 65 and over.

DETAILED DESCRIPTION:
The study is a multicenter, parallel three-group, randomized controlled study conducted to examine the effects of aerobic and resistance exercises applied within the framework of green exercise concept on physical fitness, aerobic capacity and intrinsic capacity. In this study, it was aimed to evaluate the effects of aerobic exercise and resistance exercises performed together with aerobic exercise, applied in the concept of green exercise with a multidisciplinary team (specialist doctors physiotherapists, nurses) on senior fitness, aerobic capacity and IC in individuals aged 65 and over.

ELIGIBILITY:
Inclusion Criteria:

* After the cardiology examination, it was decided that it was suitable for exercise,
* The Mini Mental Test score was above 24 points
* Had adequate communication skills

Exclusion Criteria:

* Individuals with uncontrollable arrhythmia and/or hypertension,
* neuromuscular disease,
* orthopedic injury that interferes with walking,
* severe sensory deficit, visual and/or hearing problems

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Z Score of the Intrincic Capacity | 1 week
  Z socre of the Intrincic Capacity of Elderly which calculated by tug test score, mini mental state examination score, geriatric depression scale score, mini nutritional assessement score, hand grip strength

SECONDARY OUTCOMES:
V02max | 1 week
  Aerobic Capacity of Elderly, measured by shuttle test
Senior Fitness test | 1 week
  Fitness of Elderly, measured by senior fitness test scores (higher score means better fitness level)

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Study Director — Sultan Abdülhamid Training And Research Hospital
Locations (1):
- Elif Yıldırım Ayaz, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yildirim Ayaz E, Dincer B, Mete E, Kaygusuz Benli R, Cinbaz G, Karacan E, Cankul A, Mesci B. Evaluating the impact of aerobic and resistance green exercises on the fitness, aerobic and intrinsic capacity of older individuals. Arch Gerontol Geriatr. 2024 Mar;118:105281. doi: 10.1016/j.archger.2023.105281. Epub 2023 Nov 27. PMID 38056100